CLINICAL TRIAL: NCT05918471
Title: PReoperative Very Low Energy Diets for Obese PAtients Undergoing Non-bariatric Surgery: A Randomized Evaluation (PREPARE Pilot)
Brief Title: PReoperative Very Low Energy Diets for Obese PAtients Undergoing Non-bariatric Surgery
Acronym: PREPARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Queen's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15946
Record Dates: First submitted 2023-05-18; First posted 2023-06-26 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Non-Bariatric Surgery; Preoperative Weight Loss; Preoperative Optimization
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This is a multi-center, blinded, parallel pilot RCT.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgeons, investigators, outcome assessors, and data analysts will be blinded to treatment allocation to limit measurement bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very Low Energy Diet + Standard Counselling (Experimental): All patients in the intervention group will receive standard patient counselling on weight loss and an active VLED protocol. The preoperative VLED protocol will utilize Optifast 900, a commercially available weight loss product sold by Nestlé Health Sciences. Optifast 900 is designed as a high-protein, low-carbohydrate, and low-fat meal replacement with complete micronutrient composition. Patients will receive a three-week supply. They will be instructed to consume four packets daily. This provides a total energy intake of 900 kcal. Patients will also be able to consume up to 2 cups of low-calorie vegetables per day along with the meal replacement product. They will be provided with a handout containing specific instructions. Patients will keep self-report diaries of their dietary intake and activity levels.
  Interventions: Dietary Supplement: Very Low Energy Diet with Liquid Supplementation
- Standard Counselling Alone (No Intervention): The control group patients will receive standard counselling for weight loss without prescription of a specific preoperative weight loss intervention, as this is meant to be a pragmatic trial. Currently, there are no standardized interventions aimed at optimizing obese patients prior to undergoing non-bariatric surgery. Briefly, counselling will consist of the surgeon, at the time of the preoperative clinic visit, discussing weight loss strategies such as decreased caloric intake and increased physical activity. Patients will not receive prescriptions for preoperative VLEDs, any other weight loss supplement, or any physical activity intervention aimed at promoting weight loss prior to surgery. Patients will keep self-report diaries of their dietary intake and activity levels.

INTERVENTIONS:
Dietary Supplement: Very Low Energy Diet with Liquid Supplementation — The preoperative VLED protocol will utilize Optifast 900, a commercially available weight loss product sold by Nestlé Health Sciences. Optifast 900 is designed as a high-protein, low-carbohydrate, and low-fat meal replacement with complete micronutrient composition. Instructions for use are as follows:
  1. Consume 4 Optifast 900 packets each day
  2. Take 1 sachet of Optifast 900 once in the morning (AM), once at noon, once in the early evening (PM #1), and once later in the evening (PM #2) for three-weeks.
  3. Mix 1 sachet with at least 300 mL (1 1⁄4 cups) of cold water. Shake well or blend in a blender.
  Other Names: Optifast 900
  Arms: Very Low Energy Diet + Standard Counselling

SUMMARY:
The PREPARE Pilot randomized controlled trial (RCT) is a multi-center, parallel, blinded RCT that aims to assess the feasibility of a full RCT comparing preoperative very low energy diets (VLEDs) to standard of care prior to elective non-bariatric surgery for obese patients in terms of overall 30-day postoperative morbidity. Adult patients with body mass indices (BMIs) greater than 30 kg/m2 will be randomized 1:1 to receive 3-weeks of preoperative VLED plus preoperative weight loss counselling or preoperative weight loss counselling alone. This trial will enroll patients to assess recruitment, compliance, and follow-up completion to assess the feasibility of a full RCT powered to assess for differences in 30-day postoperative between VLEDs and standard of care arms.

DETAILED DESCRIPTION:
Obesity is a worldwide epidemic affecting upwards of 700 million people. The economic burden in the United States and Canada are estimated at over $2 trillion and $100 billion United States dollars (USD), respectively, and the resultant healthcare consequences can be devastating for systems and patients alike. Obesity is a systemic disease with devastating consequences for patients undergoing any form of operative intervention. Obese patients presenting in need of medical and surgical intervention are at 2-to-6 fold higher risk of prolonged hospitalization, infectious morbidity, venous thromboembolism, and more. To pre-emptively mitigate some of these concerns, prescribed preoperative weight loss via VLEDs has become a standard of care for obese patients undergoing bariatric surgery (i.e., weight loss surgery). While VLEDs have become a standard in obese patients undergoing bariatric surgery, largely due to the significant reduction of peri-organ fat for better visualization, their application to obese patients undergoing other types of surgery remains limited. A previous systematic review and meta-analysis that identified 13 studies evaluating the use of preoperative VLEDs in obese patients undergoing orthopaedic, vascular, colorectal, upper gastrointestinal, gynecological, and a variety of general surgery procedures for benign disease (e.g., cholecystectomy, abdominal wall hernia). While data were heterogenous, preoperative VLEDs reliably resulted in significant weight loss (3.2-19.2kg) with high rates of compliance to the protocols (94-100%). Adverse event rates were low (<14% in most studies). There were no significant differences in postoperative outcomes, though again pooled analyses included a small number of patients and there were wide corresponding 95% CIs. Overall, this review suggested the evidence for routine use of VLEDs in obese patients undergoing major surgery is compromised by heterogeneous small studies with methodological limitations. A large, definitive trial is required to resolve this uncertainty. Prior to a definitive trial to compare the efficacy of VLEDs in obese patients undergoing major surgery, a pilot RCT is required. A pilot trial will provide the following critical feasibility insights: (1) Assessment of recruitment and randomization ability; (2) Evaluation of compliance to VLED regimens; and (3) Assessment of our ability follow patients completely. The objective of this pilot RCT is to determine the feasibility of a multicenter RCT comparing obese patients (i.e., BMI > 30kg/m2) receiving VLEDs versus control prior to elective non-bariatric surgery in terms of perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* BMI of greater than 30 kg/m2
* Undergoing major elective non-bariatric surgery. Major surgery is defined as any operation performed under general anesthesia requiring a skin incision extending beyond the subcutaneous tissue.

Exclusion Criteria:

* Undergoing bariatric surgery
* Undergoing neurologic surgery
* Undergoing urgent or emergent surgery
* Recently diagnosed myocardial infarction or unstable angina (i.e., within past six months)
* Diagnosed moderate-to-severe renal dysfunction (i.e., eGFR less than 30mL/min/1.73m2)
* Diagnosed severe liver dysfunction (i.e., cirrhosis, portal hypertension, hepatic encephalopathy, hepatorenal syndrome)
* Recently diagnosed alcohol or drug use disorders (i.e., excessive use of substance within past six months)
* Experienced a recent episode of gout (i.e., within past six months)
* Medical history of porphyria; (10) Known allergy to any Optifast ingredient
* Enrolled in other prospective studies with similar interventions and/or outcomes. Co-enrollment may be deemed appropriate if the steering committees of the respective trials review the details of participation.
* Pregnant or breastfeeding women
* Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  Defined as the number of patients randomized into the RCT per month.
Intervention compliance | 1 year
  Defined as the number of preoperative VLED doses taken divided by the total number of doses prescribed for each participant randomized to the intervention arm.
Follow-up completion | 1 year
  Defined as completion of the pre-VLED, preoperative, and 30-day postoperative visits, along with complete anthropometric measures and study questionnaires.
Network development | 1 year
  Defined as recruiting from all three participating centers at the aforementioned rate. Additionally, we will aim to extend our multi-disciplinary network to at least 10 centers throughout the course of this pilot RCT in preparation for the full RCT.

SECONDARY OUTCOMES:
VLED associated adverse events | Three-week VLED intervention period.
  The primary safety outcome will be all adverse events deemed secondary to the preoperative VLED. The adverse events will be recorded as dichotomous outcomes and described as either minor or serious, similarly to the OPTIWIN Study; the largest medical weight loss RCT evaluating VLEDs.
Overall 30-day postoperative morbidity | 30-days following index operation.
  This will be defined as any deviation from the usual postoperative course within 30-days of the index operation and will be a composite of system-specific complications.
30-day system-specific complications | 30-days following index operation.
  Pre-defined system-specific outcomes based on most common postoperative complications following the included types of surgery.
30-day postoperative mortality | 30-days following index operation.
  Death within 30 days of index surgery.
Preoperative weight loss | Three-week VLED intervention period.
  Preoperative weight loss will be assessed by measuring the post-VLED weight on the date of surgery and adjusting for the baseline weight in kg.
Operative time | Intraoperative
  Operative time will be measured as the time between first skin incision and closure of the last surgical wound in minutes and will be retrieved from the patient EMRs.
Intraoperative blood loss | Intraoperative
  This will be measured in milliliters and will be ascertained from the patient chart.
Surgeon-perceived technical difficulty | Intraoperative
  Surgeon-perceived difficulty will be evaluated with a short electronic questionnaire administered immediately following completion of the case.
Postoperative length of stay | Through postoperative stay, a mean of 3 days
  This will be measured in days and will be ascertained from the patient chart.
Health-related quality of life | 30 days
  Utilizing Short Form-36. The lowest and highest possible scores are 0 and 100, respectively. A higher score is associated with a greater health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler J McKechnie, MD, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - Hamilton General, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKechnie T, Ramji K, Saddik M, Leitch J, Farooq A, Patel S, Doumouras A, Parpia S, Eskicioglu C, Bhandari M. PReoperative very low-Energy diets for obese PAtients undergoing non-bariatric surgery Randomized Evaluation (PREPARE): a protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2024 May 21;10(1):82. doi: 10.1186/s40814-024-01511-6. PMID 38773543